CLINICAL TRIAL: NCT01607697
Title: Mindfulness Based Intervention (MBI) on the Quality of Life and Non-Motor Symptoms (NMS) of Persons With Parkinson's Disease (PD)
Brief Title: Mindfulness Based Intervention (MBI) on the Quality of Life and Non-Motor Symptoms (NMS) of Persons With PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr. Barbara A. Pickut, Clinical Chief Neurology and Neurorevalidation, University Hospital, Antwerp
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: B300201213369
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Training (Experimental): Group received Mindfulness Training
  Interventions: Behavioral: Mindfulness Training
- Waitlist Control (No Intervention): Group received Usual Care

INTERVENTIONS:
Behavioral: Mindfulness Training — Mindfulness Training
  Arms: Mindfulness Training

SUMMARY:
Scientific Abstract:

The investigators propose a study to examine the impact of a Mindfulness Based Intervention (MBI) on the quality of life and Non-Motor Symptoms (NMS) of persons with Parkinson's disease (PD).

NMS add significantly to the disease burden and negatively impact the quality of life in PD (1,2). In a previous study the investigators confirmed the high prevalence of NMS in PD patients with either early- or late-onset of disease (3). Despite currently available treatments, PD leads to worsening disability and there remains a need for new approaches. A Mindfulness Based Intervention may provide an important adjuvant therapy in the treatment of PD in relation to NMS and quality of life.

A minimum of 100 patients will be randomly assigned to the MBI or 'Treatment As Usual' (TAU) groups. Clinical assessments (motor and non-motor scores) will be performed in both groups. The TAU group will be offered MBI after completion of the study.

To the best of our knowledge, this is the first large scale study using MBI in this indication.

DETAILED DESCRIPTION:
The investigators propose a study to examine the impact of a Mindfulness Based Intervention (MBI) on the quality of life and Non-Motor Symptoms (NMS) of persons with Parkinson's disease (PD).

NMS add significantly to the disease burden and negatively impact the quality of life in PD (1,2). In a previous study the investigators confirmed the high prevalence of NMS in PD patients with either early- or late-onset of disease (3). Despite currently available treatments, PD leads to worsening disability and there remains a need for new approaches. A Mindfulness Based Intervention may provide an important adjuvant therapy in the treatment of PD in relation to NMS and quality of life.

A minimum of 100 patients will be randomly assigned to the MBI or 'Treatment As Usual' (TAU) groups. Clinical assessments (motor and non-motor scores) will be performed in both groups. The TAU group will be offered MBI after completion of the study.

To the best of our knowledge, this is the first large scale study using MBI in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the UK Brain Bank Criteria;
* Patients in Hoehn & Yahr stage 1-3;
* Lack of features suggestive of atypical Parkinsonism;
* No history of neuroleptics or other drugs that induce parkinsonism in the last 60 days;
* Currently optimally treated with medication and unlikely to be requiring anti-PD medication adjustments in the next 4 months;
* On a stable dose of all medications for 30 days;
* Lack of cognitive dysfunction as based on the MoCA (score ≥ 26).

Exclusion Criteria:

* Cognitive dysfunction based on the MoCA (score < 26);
* Patients with Hoehn & Yahr stage 4 and above when in 'on' stage;
* Unstable, major psychiatric or life threatening concomitant disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (PDQ-39) | 2 years

SECONDARY OUTCOMES:
Hamilton Depression Scale (Ham-D) | 2 years
MRI | 2 years
  Structural and functional MRI pre- and post-MBI

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Pickut, MD, MPH, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University Hospital Antwerp, Antwerp, Antwerp, Belgium

REFERENCES:
- [Background] Grossman P, Kappos L, Gensicke H, D'Souza M, Mohr DC, Penner IK, Steiner C. MS quality of life, depression, and fatigue improve after mindfulness training: a randomized trial. Neurology. 2010 Sep 28;75(13):1141-9. doi: 10.1212/WNL.0b013e3181f4d80d. PMID 20876468